CLINICAL TRIAL: NCT03420105
Title: Study of the Functioning of Prospective Memory in Breast Cancer and the Influence of Sleep
Acronym: PROSOM-K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PROSOM-K
Record Dates: First submitted 2018-01-10; First posted 2018-02-05 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Memory Disorders
MeSH Terms: conditions — Breast Neoplasms; Memory Disorders

STUDY DESIGN:
Intervention Model Description: 50 patients including:
  * 25 patients being treated with adjuvant hormone therapy (Group A)
  * 25 patients not receiving adjuvant hormone therapy (Group B)
  * 25 healthy volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Other): Patients perform neuropsychological, psycho-pathological and quality of life assessments, and sleep tests
  Interventions: Other: Neuropsychological, psycho-pathological and quality of life assessments; Drug: Hormonotherapy
- Group B (Other): Patients perform neuropsychological, psycho-pathological and quality of life assessments, and sleep tests
  Interventions: Other: Neuropsychological, psycho-pathological and quality of life assessments
- Healthy volunteers (Other): Healthy volunteers perform neuropsychological, psycho-pathological and quality of life assessments, and sleep tests
  Interventions: Other: Neuropsychological, psycho-pathological and quality of life assessments

INTERVENTIONS:
Other: Neuropsychological, psycho-pathological and quality of life assessments — Patients and Healthy volunteers perform neuropsychological, psycho-pathological and quality of life assessments, and sleep tests
  Other Names: sleep tests
Drug: Hormonotherapy — Adjuvant hormone therapy
  Arms: Group A

SUMMARY:
The results of this study will contribute to a better understanding of prospective memory deficit processes in breast cancer in relation to sleep disorders frequently reported in this pathology. In the long term, a better understanding will make it possible to envisage appropriate treatments to compensate for these memory difficulties and to improve the autonomy of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Major patients under the age of 70;
* Patients who have been treated by surgery or radiotherapy for non-metastatic breast cancer
* Radiotherapy completed for about 6 months
* Level of study 3 "end of primary studies" minimum (Barbizet scale);
* French mother tongue;
* Menopausal women for at least 1 year before the selection visit
* Absence of primary cancer of the central nervous system or brain metastases;
* Absence of previous neurological damage;
* Absence of personality disorders and progressive psychiatric pathology;
* Having signed the informed consent to participate in the study.

Exclusion Criteria:

* Primary cancer other than breast
* Metastatic cancer
* Treated by chemotherapy
* Cognitive function disorders pre-existing to cancer diagnosis
* Patients with paraneoplastic syndrome;
* Evolutionary psychiatric pathology;
* Refusal of participation;
* Patients unable to respond to cognitive tests;
* Drug use or excessive consumption of alcohol.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
The memory components and memory loss mechanisms by questionnaires | 6 months after the end of radiotherapy

SECONDARY OUTCOMES:
The effect of sleep quality on the recovery of intentions in prospective memory by questionnaires | 6 months after the end of radiotherapy
The impact of adjuvant hormone therapy on the functioning of prospective memory by questionnaires | 6 months after the end of radiotherapy
The influence of anxio-depressive factors and fatigue on prospective memory by questionnaires | 6 months after the end of radiotherapy

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre François Baclesse, Caen
  - Inserm-Ephe-Unicaen U1077 (, Caen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elia C, Perrier J, Duivon M, Rehel S, Gernier F, Fernette M, Doidy F, Clochon P, Grellard JM, Christy F, Segura-Djezzar C, Geffrelot J, Emile G, Allouache D, Viader F, Levy C, Joly F, Eustache F, Giffard B. Links between nocturnal hypoxia and cognitive function in breast cancer. Sci Rep. 2025 Nov 27;15(1):42405. doi: 10.1038/s41598-025-26591-z. PMID 41309988
- [Derived] Duivon M, Perrier J, Joly F, Licaj I, Grellard JM, Clarisse B, Levy C, Fleury P, Madeleine S, Lefevre N, Rauchs G, Lecouvey G, Fraisse F, Viader F, Eustache F, Desgranges B, Giffard B. Impact of breast cancer on prospective memory functioning assessed by virtual reality and influence of sleep quality and hormonal therapy: PROSOM-K study. BMC Cancer. 2018 Sep 3;18(1):866. doi: 10.1186/s12885-018-4762-2. PMID 30176833